CLINICAL TRIAL: NCT00761852
Title: Signaling Mechanisms and Vascular Function in Diabetes Mellitus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Mark A. Creager, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1999-P-003331Ruboxistaurin
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2008-09-30 (Estimated); Status verified 2008-09

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — ruboxistaurin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Ruboxistaurin
  Interventions: Drug: Ruboxistaurin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ruboxistaurin — 32 mg daily for 2 weeks
  Other Names: LY-333531
  Arms: 1
Drug: Placebo — 1 tab po QD for 2 weeks
  Arms: 2

SUMMARY:
Ruboxistaurin is being tested to see if it is effective in treating certain diabetic complications, such as diseases of the blood vessels.

DETAILED DESCRIPTION:
To test the hypothesis that activation of protein kinase C impairs vascular reactivity in patients with diabetes.

A major cause of death and disability in patients with diabetes mellitus is atherosclerosis. Endothelial dysfunction is an important, if not primary, factor in atherogenesis. Nitric oxide is an important substance made and released by the endothelium. Many prior studies in animals and humans have shown that the ability of the blood vessel to dilate is impaired in diabetes. This process of vasodilation is mediated by a substance, nitric oxide, which is thought to be highly susceptible to destruction by oxidant molecules. In previous studies, we found that acute administration of the antioxidant, vitamin C, improves endothelium-dependent vasodilation in blood vessels of patients with type 1 and type 2 diabetes. This suggests that by scavenging oxidants, such as superoxide, vitamin C may reduce the destruction of nitric oxide and thereby preserve endothelial function. Additional mechanisms, including activation of a substance called protein kinase C, and oxidant stress from excess soluble peroxides may be present in diabetes and interact with oxidant stress to cause endothelial dysfunction in patients with diabetes. Accordingly, we would like to study both of these mechanisms to determine their contribution to endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diabetes mellitus will be eligible if they are receiving dietary treatment for hyperglycemia, sulfonylureas, metformin or insulin

Exclusion Criteria:

* Any diabetic subject with a HgbA1C level of <7% or >11%
* Evidence of atherosclerosis
* symptoms of angina
* symptoms of claudication
* symptoms of cerebrovascular ischemia
* findings of arterial occlusive disease, as would be suggested by decreased pulses, asymmetric blood pressure, bruits or reduced limb pressure measurements
* hypertension defined as a systolic blood pressure > = 150 mmHg and a diastolic blood pressure >= 95 mmHg; (allowable blood pressure medications for diabetic subjects include calcium channel blockers, alpha and beta adrenergic blockers, and diuretics)
* hypercholesterolemia, defined as total cholesterol levels greater than 75th percentile for age and sex and LDL cholesterol levels >130mg/dL.
* renal insufficiency (serum creatinine >1.5 mg/dL for men; >1.2 mg/dL for women)
* hepatic dysfunction defined as liver enzyme abnormalities > two times the upper limit of normal
* chronic pulmonary disease
* congestive heart failure
* pregnancy (or subjects planning to become pregnant);
* history of cigarette smoking within the last five years;
* history of clinically significant coronary artery or cerebrovascular disease (defined as MI or stroke within 6 months, or presence of unstable angina)

  * use of any, vasoactive, cardioactive, or non-steroidal anti-inflammatory medications within 24 hours of vascular testing visits

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1999-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To test the hypothesis that activation of protein kinase Cß (PKCß) impairs vascular reactivity in patients with diabetes mellitus | one testing visit every 4 weeks for 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Creager, MD, Principal Investigator — Brigham and Women's Hospital